CLINICAL TRIAL: NCT03336593
Title: A Bridging Study to Assess Protectivity and Safety of Quadrivalent Influenza HA Vaccine in Indonesian Population
Brief Title: Protectivity and Safety of Quadrivalent Influenza HA Vaccine in Indonesian Population
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PT Bio Farma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: QIV 0217
Record Dates: First submitted 2017-11-06; First posted 2017-11-08 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-04

CONDITIONS: Safety Issues
MeSH Terms: interventions — Influenza Vaccines

STUDY DESIGN:
Intervention Model Description: Subjects 9- 40 years of age: Experimental, randomized, double blind bridging study Subjects 6 months - 8 years of age: Experimental, open labeled bridging study
Who Masked: Participant, Investigator
Masking Description: The study for subjects 9-40 years of age is randomized, double blind study. While the study for subjects 6 months-8 years of age is open labeled study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- QIV batch 1 (Experimental): 1 dose of 0.5 ml of quadrivalent influenza vaccine batch 1
  Interventions: Biological: Quadrivalent Influenza Vaccine
- QIV batch 2 (Experimental): 1 dose of 0.5 ml of quadrivalent influenza vaccine batch 2
  Interventions: Biological: Quadrivalent Influenza Vaccine
- QIV batch 3 (Experimental): 1 dose of 0.5 ml of quadrivalent influenza vaccine batch 3
  Interventions: Biological: Quadrivalent Influenza Vaccine
- Trivalent Influenza Vaccine (Active Comparator): 1 dose of 0.5 ml of trivalent influenza vaccine
  Interventions: Biological: Trivalent Influenza Vaccine
- QIV (subjects 6-35 months) (Experimental): 2 dose of 0.25 ml of quadrivalent influenza vaccine
  Interventions: Biological: Quadrivalent Influenza Vaccine
- QIV (subjects 3-8 years) (Experimental): 2 dose of 0.5 ml of quadrivalent influenza vaccine
  Interventions: Biological: Quadrivalent Influenza Vaccine

INTERVENTIONS:
Biological: Quadrivalent Influenza Vaccine — 1 or 2 doses of Quadrivalent Influenza Vaccine depends on age
  Other Names: QIV
  Arms: QIV (subjects 3-8 years); QIV (subjects 6-35 months); QIV batch 1; QIV batch 2; QIV batch 3
Biological: Trivalent Influenza Vaccine — 1 dose of Trivalent Influenza Vaccine
  Other Names: TIV
  Arms: Trivalent Influenza Vaccine

SUMMARY:
This study is to assess protectivity and safety of Quadrivalent Influenza Vaccine in Indonesian Population

DETAILED DESCRIPTION:
To describe the protectivity rate of Quadrivalent Influenza HA vaccine 28 days after immunization in Indonesian population.

To describe immunogenicity of quadrivalent Influenza HA vaccine in all subjects

ELIGIBILITY:
Inclusion Criteria for Subjects 9 - 40 Years of Age:

* Healthy
* Properly informed about the study and having signed the informed consent form
* Subject/Parent will commit themselves to comply with the instructions of the investigator and the schedule of the trial.

Inclusion Criteria for Subjects 6 Months - 8 Years of Age:

* Healthy
* Parents have been informed properly regarding the study and signed the informed consent form
* Parents will commit themselves to comply with the instructions of the investigator and the schedule of the trial

Exclusion Criteria:

* Subject concomitantly enrolled or scheduled to be enrolled in another trial
* Evolving mild, moderate or severe illness, especially infectious diseases or fever (axillary temperature >= 37.5 C )
* Known history of allergy to egg and or chicken protein or any component of the vaccines
* History of uncontrolled coagulopathy or blood disorders contraindicating intramuscular injection
* Subject who has received in the previous 4 weeks a treatment likely to alter the immune response (intravenous immunoglobulins, blood-derived products or long term corticotherapy (> 2 weeks).
* Pregnancy & Lactation (Adult)
* Any abnormality or chronic disease which according to the investigator might interfere with the assessment of the trial objectives
* Subject already immunized with influenza vaccine within 1 year.
* Subjects receive any vaccination within 1 month before and after immunization of Quadrivalent Influenza Vaccine.

Ages: 6 Months to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 810 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2018-03-14 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with an anti-influenza titer >= 1:40 HI units | 28 days after the last dose immunization
  The anti-influenza antibody serological response

SECONDARY OUTCOMES:
Geometric Mean Titer (GMT) | 28 days
  GMT in all subjects; comparison of GMT between one dose of quadrivalent and trivalent influenza HA vaccine in subjects 9-40 years old; and comparison of GMT between each batch number of quadrivalent influenza HA vaccine in subjects 9-40 years old
Percentage of subjects with increasing antibody titer >= 4 times | 28 days
  Percentage of subjects with increasing antibody titer >= 4 times: in all subjects; comparison between one dose of quadrivalent and trivalent influenza HA vaccine in subjects 9-40 years old; and comparison between each batch number of quadrivalent influenza HA vaccine in subjects 9-40 years old
Percentage of subjects with transition of seronegative to seropositive | 28 days
  Percentage of subjects with transition of seronegative to seropositive: in all subjects; comparison between one dose of quadrivalent and trivalent influenza HA vaccine in subjects 9-40 years old; and comparison between each batch number of quadrivalent influenza HA vaccine in subjects 9-40 years old
Percentage of subjects with at least one immediate reaction | 30 minutes after each vaccination
  Immediate reaction (local reaction or systemic event)
Percentage of subjects with at least one of these adverse events | within 72 hours, between 72 hours to 28 days after vaccination
  At least one of these adverse events, expected or not
Serious adverse event after vaccination | 28 days
  Serious adverse event occurring from inclusion until 28 days after vaccination.
Comparison adverse events between quadrivalent and trivalent influenza HA vaccine. | 28 days
  Adverse events occuring until 28 days after vaccination
Comparison of adverse events between each batch number of quadrivalent influenza HA vaccine. | 28 days
  Adverse events occuring until 28 days after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Meita Dhamayanti, Principal Investigator — Hasan Sadikin General Hospital
Locations (3):
- Indonesia (3):
  - Garuda Primary Health Center, Bandung, West Java
  - Ibrahim Adjie Primary Health Center, Bandung, West Java
  - Puter Primary Health Center, Bandung, West Java

REFERENCES:
- [Derived] Fadlyana E, Dhamayanti M, Tarigan R, Prodjosoewojo S, Rahmadi AR, Sari RM, Rusmil K, Kartasasmita CB. Immunogenicity and safety of Quadrivalent Influenza HA vaccine compared with Trivalent Influenza HA vaccine and evaluation of Quadrivalent Influenza HA vaccine batch-to-batch consistency in Indonesian children and adults. PLoS One. 2023 Aug 24;18(8):e0281566. doi: 10.1371/journal.pone.0281566. eCollection 2023. PMID 37616221
- [Derived] Dhamayanti M, Tarigan R, Fadlyana E, Prasetyo D, Amalia N, Rusmil VK, Sari RM, Bachtiar NS, Rusmil K, Kartasasmita CB. Immunogenicity and safety of Quadrivalent Influenza HA vaccine in Indonesian children: An open-labeled, bridging, clinical study. Vaccine. 2020 Jan 29;38(5):993-1000. doi: 10.1016/j.vaccine.2019.12.008. Epub 2019 Dec 17. PMID 31862195